CLINICAL TRIAL: NCT05127395
Title: Impact of Dosing Weight on Clinical Outcomes in Obese Patients Receiving Acyclovir for HSV Encephalitis (ID-OPRAH)
Brief Title: Impact of Obesity on Clinical Outcomes in Patients Receiving Acyclovir for HSV Encephalitis"
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 007.PHA.2020.A
Record Dates: First submitted 2021-11-09; First posted 2021-11-19 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: HSV Encephalitis
MeSH Terms: conditions — Encephalitis, Herpes Simplex

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: To assess the clinical impact of dosing acyclovir based on IBW or adjBW for HSV encephalitis to definitively guide safe and effective therapy. — The study center utilize Epic ® electronic health record (Verona, Wisconsin; www.epic.com) for which all data will be extracted from. Each study center will obtain individual IRB approval prior to data collection. SSM - St. Clare will serve as the lead center for the study with all other centers sending collected and de-identified data to this central site for analysis.

SUMMARY:
Multicenter retrospective chart review of patients admitted to any of the six study centers (SSM Health - St. Clare, St. Mary's, Saint Louis University Hospital, St. Anthony's, St. Mary's Madison, Rush University Medical Center, or Methodist Dallas Medical Center) between January 1, 2013 and December 31, 2019 will be conducted. All study centers utilize Epic ® electronic health record (Verona, Wisconsin; www.epic.com) for which all data will be extracted from. Each study center will obtain individual IRB approval prior to data collection. SSM - St. Clare will serve as the lead center for the study with all other centers sending collected and de-identified data to this central site for analysis.

DETAILED DESCRIPTION:
* Obese - WHO definition: Body Mass Index > 30 kg/m2
* Ideal Body Weight (IBW) (male) - 50.0 kg + 2.3 kg x (patient height in inches, above 60 inches)
* Ideal Body Weight (female) - 45.5 kg + 2.3 kg x (patient height inches, above 60 inches)
* Adjusted Body Weight - IBW + [0.4 x (ABW - IBW)]
* HSV encephalitis - PCR positive for HSV-1 or HSV-2 in CSF during index admission
* Baseline Serum Creatinine (S Cr) - The SCr value obtained before the start of acyclovir therapy on which the dose of acyclovir should be based upon
* Acute Kidney Injury (AKI) - per RIFLE criteria and while receiving acyclovir: SCr doubles or urine output < 0.5 mL/kg/hour for 12 hours
* End-stage renal disease (ESRD) on admission - mention of a diagnosis of ESRD in electronic medical records prior to receipt of acyclovir
* Guideline-approved, weight-based doses - within 10% of 10 mg/kg dose (to account for rounding due to vial size)
* Adequate hydration - IV fluid order (other than KVO [keep vein open]) within 24 hours before acyclovir start AND either IV fluid order (other than KVO) for majority of acyclovir course or IV fluid + oral diet for majority of acyclovir course
* Appropriately renally dose-adjusted doses - Frequency of acyclovir matches package insert recommendations based on creatinine clearance at baseline
* Interacting medications - Mycophenolate, probenecid, zidovudine, tenofovir, valproic acid, phenytoin

ELIGIBILITY:
Inclusion Criteria:

* Patients Admitted to a SSM Health - St. Clare (STL), St. Mary's (STL), Saint Louis University Hospital (STL), St. Anthony's (OKC), St. Mary's Madison (WIS), Rush University Medical Center (RUMC), or Methodist Dallas Medical Center
* > 18 years old
* Positive cerebrospinal fluid (CSF) PCR for HSV-1 or HSV-2
* BMI > 30 kg/m2
* Received guideline-approved, weight-based doses of IV acyclovir for HSV encephalitis for at least 72 hours during the index admission
* Received appropriately renal dose-adjusted doses of IV acyclovir per package insert recommendations

Exclusion Criteria:

* More than one dosing weight strategy utilized for > 24 hours for IV acyclovir dosing during the index admission
* Patients transferred to the hospital already on IV acyclovir for HSV encephalitis
* ESRD on admission
* Concomitant pathogen causing meningitis or encephalitis
* Oral acyclovir used for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * More than one dosing weight strategy utilized for > 24 hours for IV acyclovir dosing during the index admission
  * Patients transferred to the hospital already on IV acyclovir for HSV encephalitis
  * ESRD on admission
  * Concomitant pathogen causing meningitis or encephalitis
  * Oral acyclovir used for treatment
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | Over 1 month
  Will assess the clinical impact of dosing acyclovir based on IBW or adjBW for HSV encephalitis

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Crotty, PharmD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Methodist Charlton Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided